CLINICAL TRIAL: NCT00277043
Title: A Phase III Randomized Trial Assessing the Utility of a Test Dose Program With Taxanes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0902C
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2009-12

CONDITIONS: Supportive; Ill-defined Sites
Keywords: Taxane; Test Dose
MeSH Terms: interventions — Paclitaxel; Docetaxel; taxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Test Dose (Experimental)
  Interventions: Drug: paclitaxel, docetaxel, taxane
- 2) Non test dose arm (Active Comparator)
  Interventions: Drug: taxane

INTERVENTIONS:
Drug: paclitaxel, docetaxel, taxane — 1 mg paclitaxel or docetaxel test dose is prepared in 3 ml of normal saline and administered over two to five minutes IV push at least 30 minutes after prescribed IV and PO pre-medications. If no discernable adverse reaction ensues, the balance of the taxane dose is prepared and administered as per standard or specific chemotherapy protocol.
  Other Names: Taxol; Taxotere
  Arms: 1 Test Dose
Drug: taxane — The full taxane dose is prepared and administered as per standard or specific chemotherapy protocol, at least 30 minutes after prescribed IV and PO pre-medications.
  Arms: 2) Non test dose arm

SUMMARY:
The purpose of this study are to determine whether a test dose program for taxanes will reduce the rate and/or severity of hypersensitivity reactions (HSR); and to determine whether a test dose program for taxanes will result in cost reduction due to decreased drug wastage.

DETAILED DESCRIPTION:
Patients will be randomized on to one of two arms:

1. Test dose arm 1 mg paclitaxel or docetaxel test dose is prepared in 3 ml of normal saline and administered over two to five minutes IV push at least 30 minutes after prescribed IV and PO pre-medications. If no discernable adverse reaction ensues, the balance of the taxane dose is prepared and administered as per standard or specific chemotherapy protocol.
2. Non test dose arm The full taxane dose is prepared and administered as per standard or specific chemotherapy protocol, at least 30 minutes after prescribed IV and PO pre-medications.

ELIGIBILITY:
Inclusion Criteria:

* Patient must sign informed consent
* Patient must be greater than 18 years of age
* Patient must be receiving his/her first dose of either Taxol or Taxotere
* Patient must have received routine premedications for hypersensitivity reactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2002-06; Primary Completion 2004-07 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Patient HSR severity will be graded with an integer from 1 to 5 using the National Cancer Institute's Common Toxicity Criteria (CTC) for allergy/immunology. All Grade 3-4 HSRs will be reported through the FDA's MedWatch program | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States